CLINICAL TRIAL: NCT02480686
Title: Efficacy and Safety of Neutrino Therapy for Chronic HCV Genotype 1b Treatment-experienced Patients
Brief Title: Neutrino Regimen for Treatment-experienced HCV GT1 Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Humanity and Health Research Centre (Other)
Collaborators: Beijing 302 Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H&H_Neutrino Therapy
Record Dates: First submitted 2015-06-21; First posted 2015-06-24 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-08

CONDITIONS: Chronic Hepatitis C Infection
MeSH Terms: interventions — Sofosbuvir; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SOF+PEG+RBV (Experimental): Participants with HCV genotype 1b infection will receive Sofosbuvir (SOF) 400 mg +PEG+RBV for 12 weeks.
  Interventions: Drug: SOF+PEG+RBV

INTERVENTIONS:
Drug: SOF+PEG+RBV — Sofosbuvir (SOF) 400 mg tablet is administered orally once daily; Pegylated interferon alfa-2a (PEG) 180 μg was administered once weekly by subcutaneous injection; Ribavirin (RBV) was administered as a tablet orally according to body weight (< 75kg = 1000 mg and ≥ 75 kg = 1200 mg).
  Other Names: GS-7977; PSI-7977; Sovaldi®; Pegasys®; Copegus®

SUMMARY:
This study will evaluate the efficacy and safety of NEUTRINO regimen in Chinese chronic HCV genotype 1b treatment-experienced patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age equal to or greater than 18 years, with chronic genotype 1b infection;
2. HCV RNA equal to or greater than 10,000 IU/mL at Screening;
3. Cirrhosis determination;
4. Subjects who are treatment-experienced;
5. Screening laboratory values within defined thresholds;
6. Use of highly effective contraception methods if female of childbearing potential or sexually active male.

Exclusion Criteria:

1. HIV or chronic hepatitis B virus (HBV) infection;
2. Contraindications for PEG or RBV therapy;
3. Hematologic or biochemical parameters at Screening outside the protocol-specified requirements;
4. Active or recent history (≤ 1 year) of drug or alcohol abuse;
5. Hepatocellular carcinoma or other malignancy (with exception of certain resolved skin cancers);
6. Chronic use of systemic immunosuppressive agents;
7. History or current evidence of any condition, therapy, laboratory abnormality or other circumstance that might confound the results of the study, or interfere with the subject's participation for the full duration of the study, such that it is not in the best interest of the subject to participate.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-01; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with sustained virologic response 12 weeks after discontinuation of therapy (SVR12) | Post treatment Week 12
  SVR12 is defined as HCV RNA < lower limit of quantification (LLOQ) 12 weeks after last dose of study drug.
Proportion of participants with adverse events leading to permanent discontinuation of study drug(s) | Baseline up to Week 24
  Adverse events leading to permanent discontinuation of study drug(s)

SECONDARY OUTCOMES:
Change in HCV RNA From Baseline to Week 12 | Baseline up to Week 24
Proportion of participants with on-treatment virologic breakthrough and relapse | Baseline up to Week 24

CONTACTS AND LOCATIONS:
Overall Officials: George Lau, MD, Principal Investigator — Humanity and Health GI and Liver Centre; Guofeng Chen, MD, Principal Investigator — 302 Hospital
Locations (2):
- China (2):
  - Liver Fibrosis Diagnosis and Treatment Centre, 302 Hospital, Beijing, Beijing Municipality
  - Humanity and Health GI and Liver Centre, Hong Kong, Hong Kong